CLINICAL TRIAL: NCT04360993
Title: PET/CT and PET/MRI Based Treatment Modalities in the Modern Oncology
Brief Title: Role of PET/MRI in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Omar Freihat, Clinical investigator., University of Pecs
Other Study IDs: Pécs/ Oncoradiology
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer; Benign Neoplasm; Malignant Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent PET/CT & PET/MRI: Patients with head and neck cancer were underwent PET/CT and PET/MRI for staging, assessment and follow up
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Patients have received radiotherapy as a treatment modality for Head and neck cancer

SUMMARY:
Study aim was to investigate the diagnostic role of Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) in head and neck cancer.

DETAILED DESCRIPTION:
This study was assessed the role of Diffusion weighted imaging (DWI) in discriminating between benign and malignant lesions in Head and neck cancer as well as studying the relationship between glucose metabolism (18F-FDG) and Apparent diffusion coefficient (ADC) for better tumor assessment.

ELIGIBILITY:
Inclusion Criteria:

* Proved Head and neck cancer
* Underwent PET/CT and PET/MRI
* Lymph nodes due to primary Head and neck cancer.

For healthy subject:

* No previous history of malignancy.
* no inflammation or infection in the neck region.
* lymph node size <10mm.

Exclusion Criteria:

* patients treated before by radiotherapy / chemoradiotherapy
* patients underwent surgery
* artifacts

Ages: 41 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population were patients who have been diagnosed with head and neck cancer.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Difference in Apparent diffusion coefficient value between benign and malignant lesions | Baseline
  Apparent diffusion coefficient (ADC) was measured from benign and malignant lymph nodes by drawing region of interest (ROI) on the most homogeneous and most solid part in the target lymph node. Higher ADC value in Benign lymph node means that there are more water molecules movement inside the lymph node, more water molecules movement resulting in higher Apparent diffusion coefficient value. in malignant nodes and due to more tumor tissue, the result is to have lower water molecules motion so, lower ADC value.

CONTACTS AND LOCATIONS:
Overall Officials: Arpad Kovacs, MD, PhD, Study Director — University of Pecs; Cselik Zsolt, MD, PhD, Study Chair — Csolnoky Ferenc Kórház, Veszprém, Hungary; Omar Freihat, Principal Investigator — Doctoral school of health sciences, Pécs University, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Variable used in the study.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Freihat O, Toth Z, Pinter T, Kedves A, Sipos D, Cselik Z, Lippai N, Repa I, Kovacs A. Pre-treatment PET/MRI based FDG and DWI imaging parameters for predicting HPV status and tumor response to chemoradiotherapy in primary oropharyngeal squamous cell carcinoma (OPSCC). Oral Oncol. 2021 May;116:105239. doi: 10.1016/j.oraloncology.2021.105239. Epub 2021 Feb 25. PMID 33640578
- [Derived] Freihat O, Pinter T, Kedves A, Sipos D, Cselik Z, Repa I, Kovacs A. Diffusion-Weighted Imaging (DWI) derived from PET/MRI for lymph node assessment in patients with Head and Neck Squamous Cell Carcinoma (HNSCC). Cancer Imaging. 2020 Aug 8;20(1):56. doi: 10.1186/s40644-020-00334-x. PMID 32771060